CLINICAL TRIAL: NCT01104753
Title: Non-interventional Post Marketing Safety Study Confirming Efficacy and Safety of Pentasa Slow Release Tablets in Patients With Ulcerative Colitis in Common Clinical Practice
Brief Title: A Study of Pentasa in Patients With Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Other Study IDs: FE999907 CS07
Record Dates: First submitted 2010-03-26; First posted 2010-04-15 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-interventional post-authorisation safety study

SUMMARY:
Confirmation of safety profile of Pentasa slow release tablets 500 mg in patients with ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from ulcerative colitis

Exclusion Criteria:

* Hypersensitivity to mesalazine, salicylates or to any excipient
* Severe damage to liver or renal functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from ulcerative colitis
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Verify the safety profile | 1 year
  * Number of AEs/SAEs
  * Intensity and seriousness of reported AEs/SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (30):
- Czechia (30):
  - Hospital Brandýs n/Lab., Brandýs nad Labem
  - Faculty Hospital U Sv. Anny Brno, Brno
  - Hospital Břeclav, Břeclav
  - Investigational site, Chomutov
  - Hospital Chrudim, Chrudim
  - Investigational site, České Budějovice
  - Hospital Karviná, Fryštát
  - Hospital. Frýdek- Místek, Frýdek-Místek
  - Investigational site, Hodonín
  - Investigational site, Hradec Králové
  - Investigational site, Litoměřice
  - Hospitál Mladá Bolesl, Mladá Boleslav
  - Faculty Hospital Olomouc, Olomouc
  - Investigational site, Ostrava
  - Vítkovická Hospital, Ostrava
  - Gastromedic s.r.o.,ul., Pardubice
  - Faculty Hospital Bpry Plzeň, Pilsen
  - Faculty Hospital Lochotín Plzeň, Pilsen
  - Faculty Hospital Motol, Praha 5, Prague
  - NMSB, Praha 1, Prague
  - Poliklinika Prosek, Praha, Prague
  - Thomayerova hospital., Praha 4, Prague
  - VFN, Praha 2, Prague
  - ÚVN, Praha 6, Prague
  - Investigational site, Přerov
  - Hospital Svitavy, Svitavy
  - Provincial hospital, Kpt., Tábor
  - Investigational site, Ústí n.Labem
  - Hospital T. Bati Zlín, Zlín
  - Hospital Znojmo, Znojmo